CLINICAL TRIAL: NCT01723644
Title: CLINPCT Study: Clinical Reassessment Versus Procalcitonin-guided Algorithm in Order to Reduce Antibiotic Consumption in Community-acquired Pneumonia
Brief Title: Clinical Reassessment Versus Procalcitonin in Order to Shorten Antibiotic Duration in Community-acquired Pneumonia
Acronym: CLINPCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC12_0151
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Community-acquired Pneumonia
Keywords: antibiotherapy, community acquired pneumonia, procalcitonin guided guidelines, clinical reassessment
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCT guidance (Other): Group of patient " Procalcitonin " where the initiation and the stop of the antibiotic treatment are made according to a strategy guided by the PCT
  Interventions: Other: the procalcitonin arm
- clinical reassessment (Other): Group of patient where the initiation and the stop of the antibiotic treatment make following on clinical criteria and paraclinic not including the PCT.
  Interventions: Other: the clinical reassessment arm

INTERVENTIONS:
Other: the clinical reassessment arm — In the clinical reassessment arm, antibiotherapy is systematically started in the emergency department. The continuation, the discontinuation or the modification of the antibiotherapy initially prescribed in the ED were made at Day 1 and Day 5 based on clinical assessment. On Day 1, the aim of the clinical reassessment is diagnosis reassessment: to confirm or not the diagnosis of community-acquired pneumonia and to confirm or not the antibiotherapy. On Day 5, the aim of the clinical reassessment is to evaluate the possibility to stop the current antibiotherapy based on criteria for clinical stability defined by the Infectious Diseases Society of America
  Arms: clinical reassessment
Other: the procalcitonin arm — In the procalcitonin arm, initiation and discontinuation of the antibiotherapy is based on the antibiotic stewardship based on procalcitonin (PCT) cut-off ranges previously published. Re-evaluation of the clinical status and measurement of serum PCT levels is mandatory after 6-24 h in all persistently sick and hospitalized patients in who antibiotic are withheld. The PCT algorithm can be overruled by pre-specified criteria, e.g. in patients with immediately life-threatening disease. If the algorithm is overruled and antibiotics are given, an early discontinuation of antibiotic therapy after 3, 5 or 7 days is more or less endorsed based on PCT levels. In hospitalized patients with ongoing antibiotic therapy PCT levels are reassessed on days 3, 5 and 7 and antibiotics will be discontinued using the PCT cut-offs defined above.
  Arms: PCT guidance

SUMMARY:
CLINPCT study is a prospective, randomized, controlled, open intervention clinical trial including adult patients admitted in the emergency department with community-acquired pneumonia. The objective of this clinical trial is to compare two strategies: clinical reassessment and procalcitonin guided diagnostic and therapeutic strategy in patients with community-acquired pneumonia. In the clinical reassessment arm, antibiotherapy is systematically started in the emergency department. The continuation, the discontinuation or the modification of the antibiotherapy initially prescribed in the ED were made at Day 1 and Day 5 based on clinical assessment. On Day 1, the aim of the clinical reassessment is diagnosis reassessment: to confirm or not the diagnosis of community-acquired pneumonia and to confirm or not the antibiotherapy. On Day 5, the aim of the clinical reassessment is to evaluate the possibility to stop the current antibiotherapy based on criteria for clinical stability defined by the Infectious Diseases Society of America (Temperature ≤37.8°C, Heart rate ≤100 beats/min, Respiratory rate ≤24 breaths/min, Systolic blood pressure ≥90 mm Hg, Arterial oxygen saturation ≥90% or pO2 ≥60 mm Hg on room air). In the procalcitonin arm, initiation and discontinuation of the antibiotherapy is based on the antibiotic stewardship based on procalcitonin (PCT) cut-off ranges previously published. Re-evaluation of the clinical status and measurement of serum PCT levels is mandatory after 6-24 h in all persistently sick and hospitalized patients in who antibiotic are withheld. The PCT algorithm can be overruled by pre-specified criteria, e.g. in patients with immediately life-threatening disease. If the algorithm is overruled and antibiotics are given, an early discontinuation of antibiotic therapy after 3, 5 or 7 days is more or less endorsed based on PCT levels. In hospitalized patients with ongoing antibiotic therapy PCT levels are reassessed on days 3, 5 and 7 and antibiotics will be discontinued using the PCT cut-offs defined above.

ELIGIBILITY:
Inclusion criteria

* written informed consent
* age ≥ 18 years
* admittance from the community or a nursing home with the main diagnosis of community-acquired pneumonia justifying urgent antibiotherapy prescription, hospitalization for at least 6 hours after randomization and chest radiograph compatible with the diagnosis of CAP( Community acquired pneumonia )

Exclusion criteria

* the inability to give written informed consent
* hospitalization >24 hours
* aspiration pneumonia
* nosocomial pneumonia
* purulent pleurisy
* exacerbation of COPD (chronic obstructive pulmonary disease)
* neutropenia (<1G/L cells)
* chronic infection with current antibiotherapy
* antibiotherapy before admission for the current infection
* immunosuppression (including prolonged corticotherapy (10 mg of prednisone per day for at least one month)
* active neoplastic disease, organ transplant, pregnancy, HIV diagnosis with a CD4 count<200 cells/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
duration of antibiotic therapy expressed in days of therapy | Between Day 1 and Day 30
  antibiotic duration is defined as all antibiotherapy prescribed for a community acquired pneumonia during the 30 day following period Safety Issue: Yes

SECONDARY OUTCOMES:
clinical success at Day 30 | Day 30
  clinical success is defined as cure of the pneumonia at Day 30 Safety Issue: Clinical cure was defined as either the return to the pre-infection state (i.e. all pneumonia-related signs and symptoms had disappeared and chest X-ray findings had shown improvement) or improvement in related post-infectious stigmata, such that residual symptoms if any did not require additional treatment and were accompanied by improvement or lack of progression based on chest X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Montassier, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - University hospital of Agen, Agen
  - University Hospital of Angers, Angers
  - University Hospital of Brest, Brest
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - University Hospital of Lille, Lille
  - CHU de Nantes, Nantes
  - University Hospital of Bichat Paris, Paris
  - University Hospital of Bobigny Paris, Paris
  - University Hospital of Hôtel-Dieu Paris, Paris
  - University Hospital of Saint Antoine Paris, Paris
  - University Hospital of Rennes, Rennes
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Tours, Tours

REFERENCES:
- [Derived] Montassier E, Javaudin F, Moustafa F, Nandjou D, Maignan M, Hardouin JB, Annoot C, Ogielska M, Orer PL, Schotte T, Bouget J, Agha Babaei S, Raynal PA, Eche A, Duc AT, Cojocaru RA, Benaouicha N, Potel G, Batard E, Talan DA. Guideline-Based Clinical Assessment Versus Procalcitonin-Guided Antibiotic Use in Pneumonia: A Pragmatic Randomized Trial. Ann Emerg Med. 2019 Oct;74(4):580-591. doi: 10.1016/j.annemergmed.2019.02.025. Epub 2019 Apr 11. PMID 30982631